CLINICAL TRIAL: NCT05270018
Title: Effect of Bacterial Lysates on Respiratory Tract Microecology in Patients With Mechanical Ventilation and Evaluation of the Efficacy of Prevention and Treatment of Ventilator-associated Pneumonia
Brief Title: Bacterial Lysates on Respiratory Tract Microecology and Evaluation of the Efficacy of Prevention and Treatment of VAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheng Wang MD PhD (Other)
Responsible Party: Sponsor-Investigator, Sheng Wang MD PhD, Director, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STPH-ICU-005
Record Dates: First submitted 2021-12-29; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Ventilators, Mechanical
Keywords: Ventilators; Bacterial Lysates; Microecology; pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Bacterial Lysates; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacterial Lysate group (Experimental): Oral / gastric administration of bacterial lysate once a day on an empty stomach, 14.0mg each time for at least 5 days
  Interventions: Drug: Bacterial Lysates
- Control group (Placebo Comparator): Oral / gastric administration of normal saline once a day, 14.0ml each time
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: Bacterial Lysates — 14mg once a day
  Other Names: Fan fusu
  Arms: Bacterial Lysate group
Other: normal saline — 14.0ml once a day
  Arms: Control group

SUMMARY:
The purpose of this study is to assess the effect of bacterial lysates on respiratory tract microecology in patients with mechanical ventilation and the efficacy of prevention and treatment of ventilator associated pneumonia.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a one-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner in a 1:1 ratio to Bacterial Lysates( 14mg, once a day) or placebo(once a day).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU for mechanical ventilation
* The expected mechanical ventilation time is more than 72h
* Sign the informed consent form when conscious and voluntary, and complete the questionnaire survey and follow-up as required; If it is unable to sign the informed consent form and complete the questionnaire survey and follow-up, the legal representative or guardian can act on behalf of it.

Exclusion Criteria:

* Ventilator associated pneumonia is known and confirmed
* Pregnant or lactating female
* Allergic to the active ingredients of bacterial lysates or any excipients listed in the ingredients
* Patients with autoimmune diseases
* Patients with acute intestinal infection
* Patients participating in other clinical studies at the same time
* Patients considered unsuitable by other researchers to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
VAP incidence | 2 weeks
  The incidence rate of ventilator associated pneumonia

SECONDARY OUTCOMES:
Assessment of human immune status | one week
  Immune status Assessment of IgG, IgA, and IgM levels Quantifications of IgG, IgA, and IgM levels were determined by Immunological Turbidity Kits
drug resistant bacteria Incidence | one week
  The incidence rate of drug resistant bacteria
Composition of respiratory bacteria | one week
  probiotics and pathogens via NGS analysis
survival rate | 28 days
  ICU in-hospital mortality and 28 day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China